CLINICAL TRIAL: NCT06382181
Title: A Multimodal Intervention for Community-dwelling Individuals With Unwanted Loneliness: Music Therapy, Health Education, and Physical Exercise
Brief Title: A Multimodal Intervention for Community-dwelling Individuals With Unwanted Loneliness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, María-Vanesa Ibáñez-del-Valle, Principal Investigator, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023- ENFPOD-2621979; Silvia Corchón Arreche (Other: University of Valencia); Omar Cauli (Other: University of Valencia)
Record Dates: First submitted 2024-04-08; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Loneliness; Mental Health Disorder
Keywords: Music Therapy
MeSH Terms: conditions — Mental Disorders | interventions — Music Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: Participants were assigned to three groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Therapy (Experimental): Through listening to songs, singing, dancing, guided relaxation with music and instrumental group performance, the enjoyment and expression of feelings will be encouraged.
  Interventions: Behavioral: Music therapy for community-dwelling individuals with unwanted loneliness
- Health education (Experimental): Health education workshops
  Interventions: Behavioral: Health education for community-dwelling individuals with unwanted loneliness
- Physical exercise (Experimental): Physical exercise adapted to the physical conditions of each participant
  Interventions: Behavioral: Physical exercise for community-dwelling individuals with unwanted loneliness

INTERVENTIONS:
Behavioral: Music therapy for community-dwelling individuals with unwanted loneliness — Music therapy workshops were implemented. The enjoyment and expression of feelings were encouraged by listening to songs, singing, dancing, guided relaxation with music, and group instrumental performance. There was one session per week. Total 12 sessions.
  Other Names: Music therapy
  Arms: Music Therapy
Behavioral: Health education for community-dwelling individuals with unwanted loneliness — Twelve health education workshops were carried out. They included group training talks on the following topics: sleep hygiene, diet, and cognitive stimulation, among others.
  Other Names: Health education
  Arms: Health education
Behavioral: Physical exercise for community-dwelling individuals with unwanted loneliness — This intervention was implemented with 2 group sessions each week for 13 weeks. It included physical exercise adapted to the physical conditions of each participant.
  Other Names: Physical exercise
  Arms: Physical exercise

SUMMARY:
The absence of social relationships negatively affects physical, psychological, and social health. In other words, it alters people's quality of life and makes active aging difficult. The investigators have designed a study to reduce unwanted loneliness in people over 65 living in the community through multiple interventions (music therapy, health education, and physical exercise).

DETAILED DESCRIPTION:
The proposed study will involve 4 group sessions each week for a total of 13 weeks. The program will include the following activities:

Physical exercise adapted to the physical conditions of each participant. Total of 26 sessions (2 per week).

Health education workshops. A total of 12 workshops. These will include group training talks on the following topics: sleep hygiene, diet, and cognitive stimulation, among others.

Music therapy workshops. Through listening to songs, singing, dancing, guided relaxation with music, and group instrumental performance, the enjoyment and expression of feelings will be encouraged. There will be 1 session per week. Total 12 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Over 60 years of age with unwanted loneliness
* Must live in the city of Valencia
* Must speak Spanish or Valencian (or have sufficient knowledge to be able to answer the questions in the study).

Exclusion Criteria:

+ Severe mental disorder or dementia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Score on the Jong Gierveld Loneliness Scale | 3 months
  Social isolation was measured with the Jong Gierveld Loneliness Scale.
  The final score is the total score for the 11 items, with the lowest possible score being 0 (no loneliness) and the highest being 11 (severe loneliness). Three categories have been proposed based on the score: a score of 0-2 points = no loneliness; a score of 3-8 points = moderate loneliness; and a score of 9-11 points = severe loneliness.

SECONDARY OUTCOMES:
Score on Goldberg Anxiety and Depression Scale | 3 months
  The symptoms of anxiety and depression were measured with the Goldberg Anxiety and Depression Scale.
  This is a questionnaire that discriminates between the diagnosis of anxiety and depression and measures their retrospective intensities. It consists of two subscales: one for anxiety and one for depression. Each subscale is composed of 9 dichotomous response items (YES or NO) to determine whether the subject has had any of the indicated symptoms in the last two weeks. The cut-off points are 4 or more items or affirmative responses for the anxiety scale and 2 or more for the depression scale. The higher the score, the greater the severity of the problem, with a maximum possible score of 9 points for each subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Ibáñez del Valle, PhD, Principal Investigator — University of Valencia
Locations (2):
- Spain (2):
  - University of Valencia, Valencia
  - Vanessa Ibáñez del Valle, Valencia

IPD SHARING:
Plan to Share IPD: No
Results are expected to be shared through scientific articles in peer-reviewed journals.

REFERENCES:
- [Derived] Mafla-Espana MA, Corchon S, Jimeno-de Pedro P, Ibanez-Del Valle V, Cauli O. Social and Mental Health Factors Involved in the Severity of Loneliness in Older Individuals in a Spanish Rural Area. Nurs Rep. 2024 Nov 29;14(4):3737-3753. doi: 10.3390/nursrep14040273. PMID 39728634